CLINICAL TRIAL: NCT01539603
Title: Comparison of Drug-Eluting Balloon First and Then Bare Metal Stent With Drug-eluting Stent for Treatment of de Novo Lesions (DEB First): A Randomized Controlled Single Center Clinical Trial
Brief Title: Comparison of Drug Eluting Balloon and Drug Eluting Stent
Acronym: DEBfirst
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hwan Yoon, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-1104/061-001
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina; NSTEMI
Keywords: drug eluting balloon; bare metal stent; drug eluting stent; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB-BMS (Experimental): Drug eluting balloon + Bare metal stent
  Interventions: Device: Drug eluting balloon + Bare metal stent
- Drug eluting stent (Active Comparator): conventional PCI with drug eluting stent drug eluting stent (Zotarolimus-eluting stent)
  Interventions: Device: drug eluting stent (Zotarolimus-eluting stent)

INTERVENTIONS:
Device: Drug eluting balloon + Bare metal stent — PCI using Sequent Please and then Coroflex Blue
  Other Names: Sequent Please (B.Braun, drug eluting balloon); Coroflex Blue (B.Braun, bare metal stent)
  Arms: DEB-BMS
Device: drug eluting stent (Zotarolimus-eluting stent) — conventional PCI using Endeavor Integrity
  Other Names: Endeavor integrity; Zotarolimus-eluting stent
  Arms: Drug eluting stent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Drug-Eluting Balloon first and then bare metal stent compared with drug-eluting stent for treatment of de novo lesions (DEB first).

DETAILED DESCRIPTION:
A recent trial to test premount bare metal stent on drug-eluting balloon failed to demonstrate non-inferiority and safety compared to drug-eluting stent alone for treatment of coronary artery stenosis.

We think that inappropriate drug delivery to diseased vessel due to stent strut might affect the efficacy of drug-eluting balloon. Therefore, we design a clinical study with a different protocol, that is, drug-eluting balloon first and then bare metal stent implantation in comparison to drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesion
* 2.5mm =< Reference diameter =< 4mm
* Lesion length =< 28mm
* Type A, B1/B2 lesion

Exclusion Criteria:

* ST-segment elevation MI
* Reference diameter < 2.5mm or > 4mm
* Bifurcation lesion
* Type C lesion
* history of AMI or stroke within 1 year F. chronic renal disease (Cr > 2mg/dL)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
in-segment late loss | 9 month
  angiographic in-segment late loss measure by QCA program

SECONDARY OUTCOMES:
stent thrombosis | 9 month
  any stent thrombosis
angiographic and procedure success | 9 month
  Angiographic success denotes that residual diameter stenosis is less than 10% without complication such as coronarhy dissection or thrombosis.
  Procedural success means that adequate DEB+BMS or DES delivery to the target lesion without geographic miss.
MACE | 9 month
  death, MI and TVF

CONTACTS AND LOCATIONS:
Overall Officials: In-Ho Chae, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Universtiy Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Chae IH, Yoon CH, Park JJ, Oh IY, Suh JW, Cho YS, Youn TJ, Choi DJ. Comparison of Drug-Eluting Balloon Followed by Bare Metal Stent with Drug-Eluting Stent for Treatment of de Novo Lesions: Randomized, Controlled, Single-Center Clinical Trial. J Korean Med Sci. 2017 Jun;32(6):933-941. doi: 10.3346/jkms.2017.32.6.933. PMID 28480650
- [Derived] Park SD, Yoon CH, Oh IY, Suh JW, Cho YS, Youn TJ, Choi DJ, Chae IH. Comparison of a drug-eluting balloon first and then bare metal stent with a drug-eluting stent for treatment of de novo lesions: study protocol of a randomized controlled trial. Trials. 2013 Feb 8;14:38. doi: 10.1186/1745-6215-14-38. PMID 23394404